CLINICAL TRIAL: NCT06935435
Title: Effects of Distinct Nebraska-Dry Bean Market Classes on Gut Microbiota
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska Lincoln (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: UNL-00024307
Record Dates: First submitted 2025-03-13; First posted 2025-04-20 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Dietary Intervention; Gut Microbiota
Keywords: Dry Beans; Gut Microbiota; Nutritional Microbiology

STUDY DESIGN:
Intervention Model Description: The study intervention will consist of individuals consuming daily, precooked and prepackaged dry beans over three 2-week intervention periods. The amount of beans to consume will be ½ cups/day during week 1 and 1 ½ cups/day during week 2. The three bean interventions will be i) pink beans, ii) great northern beans, and iii) a five-bean mixture (pinto, kidney, black, pink, and great northern beans). The participants will be asked to consume all bean interventions in random order. The beans will be added to the participants' usual diet.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Intervention Scheme 1 (Active Comparator): Intervention Phase 1: Week 1: ½ cup Pink Bean → Week 2: 1½ cups Pink Bean Intervention Phase 2: Week 1: ½ cup Great Northern Bean → Week 2: 1½ cups Great Northern Bean Intervention Phase 3: Week 1: ½ cup Bean Mix → Week 2: 1½ cups Bean Mix
  Interventions: Other: Pink Beans; Other: Great Northern Beans; Other: Five-Bean Mixture
- Intervention Scheme 2 (Active Comparator): Intervention Phase 1: Week 1: ½ cup Great Northern Bean → Week 2: 1½ cups Great Northern Bean Intervention Phase 2: Week 1: ½ cup Bean Mix → Week 2: 1½ cups Bean Mix Intervention Phase 3: Week 1: ½ cup Pink Bean → Week 2: 1½ cups Pink Bean
  Interventions: Other: Pink Beans; Other: Great Northern Beans; Other: Five-Bean Mixture
- Intervention Scheme 3 (Active Comparator): Intervention Phase 1: Week 1: ½ cup Bean Mix → Week 2: 1½ cups Bean Mix Intervention Phase 2: Week 1: ½ cup Pink Bean → Week 2: 1½ cups Pink Bean Intervention Phase 3: Week 1: ½ cup Great Northern Bean → Week 2: 1½ cups Great Northern Bean
  Interventions: Other: Pink Beans; Other: Great Northern Beans; Other: Five-Bean Mixture
- Intervention Scheme 4 (Active Comparator): Intervention Phase 1: Week 1: ½ cup Pink Bean → Week 2: 1½ cups Pink Bean Intervention Phase 2: Week 1: ½ cup Bean Mix → Week 2: 1½ cups Bean Mix Intervention Phase 3: Week 1: ½ cup Great Northern Bean → Week 2: 1½ cups Great Northern Bean
  Interventions: Other: Pink Beans; Other: Great Northern Beans; Other: Five-Bean Mixture
- Intervention Scheme 5 (Active Comparator): Intervention Phase 1: Week 1: ½ cup Great Northern Bean → Week 2: 1½ cups Great Northern Bean Intervention Phase 2: Week 1: ½ cup Pink Bean → Week 2: 1½ cups Pink Bean Intervention Phase 3: Week 1: ½ cup Bean Mix → Week 2: 1½ cups Bean Mix
  Interventions: Other: Pink Beans; Other: Great Northern Beans; Other: Five-Bean Mixture
- Intervention Scheme 6 (Active Comparator): Intervention Phase 1: Week 1: ½ cup Bean Mix → Week 2: 1½ cups Bean Mix Intervention Phase 2: Week 1: ½ cup Great Northern Bean → Week 2: 1½ cups Great Northern Bean Intervention Phase 3: Week 1: ½ cup Pink Bean → Week 2: 1½ cups Pink Bean
  Interventions: Other: Pink Beans; Other: Great Northern Beans; Other: Five-Bean Mixture

INTERVENTIONS:
Other: Pink Beans — Pink beans consumed for 2 weeks, at an amount of ½ cup/day for week 1 and 1 ½ cups/day for week 2.
Other: Great Northern Beans — Great northern beans consumed for 2 weeks, at an amount of ½ cup/day for week 1 and 1 ½ cups/day for week 2.
Other: Five-Bean Mixture — Five-bean mixture made of pinto, kidney, black, pink, and great northern beans consumed for 2 weeks, at an amount of ½ cup/day for week 1 and 1 ½ cups/day for week 2.

SUMMARY:
Beans are well known for their health benefits. Many of these benefits relate to gut health, as many of the nutrients found in beans support beneficial microbes that live in the gut. However, beans have a lot of genetic diversity. This diversity has led to different bean market classes with different colors, sizes, and nutrient profiles. Differences between bean market classes may trigger different effects on gut microbes and health, but this is poorly understood. The goal of the pilot clinical trial is to make comparisons (1) between two different bean market classes (pink beans, great northern beans) and (2) between a bean mixture (pinto, kidney, black, pink, and great northern beans) and individual bean market classes. The study will assess whether bean market classes differ in their effects on gut microbes, blood pressure, metabolism, and gut symptoms in adults with and without obesity.

DETAILED DESCRIPTION:
Bean consumption delivers diverse dietary fibers (resistant starches, non-starch polysaccharides), proteins, polyphenols, and other compounds to the colon, where they serve as substrates for the microbial community (microbiota) that colonizes the gut of humans. However, dry beans exhibit high genetic diversity, corresponding with diverse pigments and nutrients across market classes. It remains poorly understood whether targeted effects on the gut microbiota and health measures are possible with distinct dry bean market classes. The overarching study objective is to perform a randomized, crossover pilot intervention trial in adults to determine the effects of consuming distinct dry bean market classes in isolation or combination on the gut microbiota and health. The study will compare the dose-dependent effects of pink beans, great northern beans, and a five-bean mixture (pinto, kidney, black, pink, and great northern beans) on the gut microbiota, health-relevant metabolites, blood pressure, and immunometabolic markers in adults with and without extra body weight. The pilot study will employ a 3-phase, cross-over design with 2-week intervention periods separated by 2-week washout periods.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 19 to 50 years.
2. Not currently pregnant or planning to become pregnant (Females Only).
3. Stable body mass index (BMI) of either 18.5-24.9 kg/m2 or 27.0-39.9 kg/m2 for the last month.
4. Has not made any major dietary changes in the last month.
5. Able to read and speak English
6. Requires no legally authorized representative (LAR).
7. Not institutionalized (e.g., prison, psychological treatment center, etc.).
8. Able to wear ambulatory blood pressure monitor and limit physical activity over a 24-hr. period.
9. Have a bowel movement at least every other day.
10. Able to collect and deliver stool samples to Innovation Campus within 4 hours of collection.
11. No known allergies or intolerance to beans.
12. Able to avoid consuming beans during the study, except for the provided beans (up to 1.5 cups/day).

Exclusion Criteria:

1. Has a cardiac device.
2. History of organ transplant
3. History of gastrointestinal surgery or disease diagnosed by a physician that involves the stomach, small, and large intestines (e.g., IBD, IBS, chronic constipation, diverticulosis, gastric bypass).
4. Recent history of cancer (excluding skin cancer) in the last year.
5. Current use of tobacco or vaping.
6. Current or recent use (last 3 weeks) of digestive enzymes, laxatives, dietary fiber, prebiotic, or probiotic supplements.
7. Medication or supplement regimen or dosage changed within the last 2 months or 3 weeks, respectively.
8. Taken antibiotics in the last 2 months.
9. Known allergies or intolerances to beans.
10. BMI 18.5-24.9 kg/m2 (normoweight): Current use of oral or injectable medications for the treatment of most chronic conditions.
11. BMI 27.0-39.9 kg/m2 (overweight): Current use of oral or injectable medications for the treatment of diabetes, hypertension, cardiovascular, liver, kidney, gastrointestinal, or autoimmune.

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-05-08 (Actual); Primary Completion 2026-01-28 (Actual); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
16S rRNA gene amplicon sequencing of the fecal bacterial community | From baseline to end of weeks 1 and 2 of treatment.
  Dose-dependent changes in bacterial composition, and precisely the relative abundance of Faecalibacterium, in fecal samples, as assessed by 16S rRNA gene amplicon sequencing.

SECONDARY OUTCOMES:
Fecal short-chain fatty acids assessed by gas chromatography | From baseline to end of weeks 1 and 2 of treatment.
  Dose-dependent changes in fecal concentrations of short-chain fatty acids as determined by gas chromatography.
Gastrointestinal symptoms assessed by the Gastrointestinal Symptom Rating Scale | From baseline to end of weeks 1 and 2 of treatment.
  Dose-dependent changes in gastrointestinal symptoms as assessed by the Gastrointestinal Symptom Rating Scale, where the scale is between 0 and 6 and higher values indicate more severe gastrointestinal symptoms.
Bowel movement habits assessed by a Bowel Habits Questionnaire | From baseline to end of weeks 1 and 2 of treatment.
  Dose-dependent changes in bowel movement (BM) habits as assessed using a Bowel Habits Questionnaire, which has been previously described by Deehan and colleagues. The questionnaire asks participants to record and describe their BMs over three-days to obtain information on BM frequency (number of BM/day), stool consistency (Bristol Stool Scale, 1 [hard] to 7 [liquid]), perceived stool hardness (1 [soft] to 4 [very hard]), straining during bowel movement, discomfort during bowel movement, sensation of incomplete evacuation (1 [none] to 4 [severe]).

OTHER OUTCOMES:
Blood pressure | From baseline to the end of treatment at 2 weeks.
  Changes in 24-hour blood pressure as evaluated by an ambulatory blood pressure monitor.
Systematic inflammation assessed by C-reactive protein | From baseline to the end of treatment at 2 weeks.
  Changes in circulating levels of C-reactive protein (Unit: mg/L) when collected after fasting.
Systematic inflammation assessed by glycosylated acute-phase proteins (GlycA) | From baseline to the end of treatment at 2 weeks.
  Changes in circulating levels of glycosylated acute-phase proteins (Unit: umol/L) when collected after fasting.
Glucose metabolism assessed by Homeostasis Model Assessment of Insulin Resistance (HOMA-IR) | From baseline to the end of treatment at 2 weeks.
  Changes in circulating levels of glucose (Unit: mg/dL) and insulin (Unit: uIU/mL) when collected after fasting. Glucose and insulin values will then be used to calculate the Homeostasis Model Assessment of Insulin Resistance using the equation previously described by Matthews and colleagues.
Glucose metabolism assessed by C-peptide | From baseline to the end of treatment at 2 weeks.
  Changes in circulating levels of C-peptide (Unit: ng/mL) when collected after fasting.
Lipid metabolism assessed by a lipid panel | From baseline to the end of treatment at 2 weeks.
  Changes in circulating levels of total cholesterol, high-density lipoprotein, low-density lipoprotein, and triglycerides (Units: mg/dL) when collected after fasting.
Percent body fat assessed by bioelectrical impedance analysis | From baseline to the end of treatment at 2 weeks.
  Changes in percent body fat assessed by an InBody 770 bioelectrical impedance analyzer. The validity of the InBody 770 bioelectrical impedance analyzer has been previously described by Brewer and colleagues.

CONTACTS AND LOCATIONS:
Overall Officials: Edward C Deehan, PhD, RD, Principal Investigator — University of Nebraska Lincoln
Locations (1):
- Nebraska Food for Health Center, Lincoln, Nebraska, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified gut bacteria sequencing data, along with limited participant information, will be uploaded to the National Center for Biotechnology Information Sequence Read Archive.
Time Frame: The de-identified gut bacteria sequencing data will be made available upon publication of study findings.
Access Criteria: Data will be available for download at the National Center for Biotechnology Information Sequence Read Archive.
URL: https://www.ncbi.nlm.nih.gov/sra

REFERENCES:
- [Background] Deehan EC, Yang C, Perez-Munoz ME, Nguyen NK, Cheng CC, Triador L, Zhang Z, Bakal JA, Walter J. Precision Microbiome Modulation with Discrete Dietary Fiber Structures Directs Short-Chain Fatty Acid Production. Cell Host Microbe. 2020 Mar 11;27(3):389-404.e6. doi: 10.1016/j.chom.2020.01.006. Epub 2020 Jan 30. PMID 32004499
- [Background] Brewer GJ, Blue MNM, Hirsch KR, Saylor HE, Gould LM, Nelson AG, Smith-Ryan AE. Validation of InBody 770 bioelectrical impedance analysis compared to a four-compartment model criterion in young adults. Clin Physiol Funct Imaging. 2021 Jul;41(4):317-325. doi: 10.1111/cpf.12700. Epub 2021 Apr 1. PMID 33752260
- [Background] Matthews DR, Hosker JP, Rudenski AS, Naylor BA, Treacher DF, Turner RC. Homeostasis model assessment: insulin resistance and beta-cell function from fasting plasma glucose and insulin concentrations in man. Diabetologia. 1985 Jul;28(7):412-9. doi: 10.1007/BF00280883. PMID 3899825

DOCUMENTS (1):
  • Informed Consent Form (2025-02-14): https://cdn.clinicaltrials.gov/large-docs/35/NCT06935435/ICF_000.pdf